CLINICAL TRIAL: NCT00483171
Title: A 14-Month, Randomized, Double-Blind,Placebo-Controlled Phase 3 Study To Evaluate The Long-Term Efficacy And Safety of CP-945,598 In Prevention Of Weight Regain In Obese Subjects
Brief Title: A 14-Month Study On The Effects Of CP-945,598 For The Prevention Of Weight Regain In Obese Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5351028
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: CP-945,598
- Non-pharmacological weight loss program (NPP) (Other)
  Interventions: Behavioral: Non-pharmacological weight loss program (NPP)
- Low Calorie Diet (Other)
  Interventions: Behavioral: Low Calorie Diet

INTERVENTIONS:
Drug: CP-945,598 — CP-945,598
  Arms: Placebo
Behavioral: Non-pharmacological weight loss program (NPP) — Nutrition counseling, exercise monitoring and behavioral management will occur for all arms during the NPP.
  Arms: Non-pharmacological weight loss program (NPP)
Behavioral: Low Calorie Diet — Low calorie diet
  Arms: Low Calorie Diet

SUMMARY:
The purpose of this study is to determine if CP-945,598 is effective in the prevention of weight regain in obese subjects.

DETAILED DESCRIPTION:
The CP-945,598 program was terminated on November 3, 2008 due to changing regulatory perspectives on the risk/benefit profile of the CB1 class and likely new regulatory requirements for approval. No safety issues were involved in the termination decision.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be overweight (BMI) >/=30 kg/m2, for subjects without co morbidities; >/=27 kg/m2 for subjects with co morbidities
* Subjects who are willing and able to comply with 8 week Low Calorie Diet, scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Participation in a formal weight loss program or significant weight loss (fluctuation >5% of total body weight) in the past 3 months.
* Subjects with serious medical or psychiatric conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Percent weight regained during the 12 month treatment period after a prior weight loss on the low calorie diet (8 weeks). | 14 months

SECONDARY OUTCOMES:
To explore the effect of CP 954, 598 on: Waist circumference | 14 months
To evaluate the safety and tolerability of CP 945,598 urine and blood tests | 14 months
To explore the effect of CP 954, 598 on: Pharmacodynamic measurements including fasting insulin, fasting plasma glucose, adiponectin | 14 months
To explore the effect of CP 954, 598 on: Patient reported outcomes: Power of Food Scale and Three factor Eating Scale | 14 months
To explore the effect of CP 954, 598 GAD 7 and PHQ 9 self report questionnaires. and C-SSRS semi structured interview | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (9):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Seattle, Washington
- Australia (5):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Kippa-Ring, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Heidelberg, Victoria
- Denmark (4):
  - Pfizer Investigational Site, Aarhus
  - Pfizer Investigational Site, Frederiksberg C
  - Pfizer Investigational Site, Gentofte Municipality
  - Pfizer Investigational Site, Roskilde
- Netherlands (3):
  - Pfizer Investigational Site, Almere Stad
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Hilversum
- South Africa (4):
  - Pfizer Investigational Site, Cape Town, Gauteng
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Pretoria

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351028&StudyName=A%2014-Month%20Study%20On%20The%20Effects%20Of%20CP-945%2C598%20For%20The%20Prevention%20Of%20Weight%20Regain%20In%20Obese%20Patients